CLINICAL TRIAL: NCT02368600
Title: A Randomized Controlled Trial Examining the Effectiveness of a Lifestyle Intervention in Reducing Gestational Diabetes Mellitus in High Risk Chinese Pregnant Women in Hong Kong
Brief Title: Lifestyle Intervention and Prevention of Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ruth Chan, Research assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014.373-T
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Gestational Diabetes Mellitus
Keywords: lifestyle intervention; gestational diabetes mellitus; Chinese; prevention
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle modification program (Experimental): On top of the usual care, subjects in the intervention will receive a lifestyle intervention that will be delivered by experienced registered dietitian and exercise specialist. There will be 5 face-to-face dietitian consultations, 2 telephone dietitian consultations and at least one face-to-face exercise specialist consultation. The exercise consultation will be normally scheduled on the same day of the face-to-face dietitian consultation.
  Interventions: Behavioral: Lifestyle modification program
- Usual care (No Intervention): Women will have their first AN booking visit generally on or before 12 week gestation. For women who are primigravida, their AN visit appointments will be set at every 6 weeks before 24 weeks, every 4 weeks between 24-28 weeks, and every 2 weeks after 28 weeks. For women who are multigravida, the corresponding schedules will be set at every 6 weeks before 24 weeks, every 4 weeks between 24-36 weeks, and every 2 weeks after 36 weeks. Body weight of the pregnant woman will be monitored by nurses and basic nutrition advice will be briefly given by nurses in case she is slightly overweight. They will be provided with an educational pamphlet on diet and exercise during pregnancy. They will also be offered optional antenatal classes which subjected to quotas availability.

INTERVENTIONS:
Behavioral: Lifestyle modification program — On top of the usual care, subjects in the intervention will receive a lifestyle intervention that will be delivered by experienced registered dietitian and exercise specialist. There will be 5 face-to-face dietitian consultations, 2 telephone dietitian consultations and at least one face-to-face exercise specialist consultation. The exercise consultation will be normally scheduled on the same day of the face-to-face dietitian consultation.
  Arms: Lifestyle modification program

SUMMARY:
The number of women with gestational diabetes mellitus (GDM) had been increasing. Maternal GDM has a great impact on both the health of the mothers and the offspring. Antenatal lifestyle interventions, in particular dietary intervention appear to be feasible to improve maternal GDM and weight gain. To the best of our knowledge, there has been no such trial examining the feasibility of a lifestyle intervention in pregnant women in Hong Kong. Therefore, we plan to conduct a randomized controlled trial comparing a lifestyle modification program (LMP) in early pregnancy and the usual antenatal care in high risk Chinese pregnant women in Hong Kong. Intervention group subjects (n=110) will participate in a dietitian-led LMP including dietary and exercise component from the first antenatal (AN) booking to 24 weeks gestation. 110 women in the control group will receive routine hospital antenatal care. The primary endpoint will be the prevalence of GDM measured using a 75 g oral glucose tolerance test at 24-28 weeks gestation. The secondary endpoints will be the proportion of infant born with large for gestational age (>=95th percentile of the customized birth weight) and macrosomia (>=4 kg at birth). The intervention group involves dietary and exercise advice and monitoring. No drug or invasive procedure is involved. The control group will receive routine antenatal care and will be provided with an educational pamphlet on diet and exercise during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin
* Reside normally in Hong Kong
* Singleton pregnancy
* Gestational age <= 12 weeks at the time of recruitment
* Could speak and understand Chinese
* Fulfill at least one of the following criteria for high risk of GDM at the time of recruitment based on the update hospital protocol implemented since 1st May 2014
* Maternal age >= 35 years old at expected date of confinement.
* Prior history of GDM or birth of child >= 4 kg
* Pre-pregnant BMI or BMI at 1st trimester >= 25 kg/m2
* Family history of diabetes at 1st degree relatives
* Willing to give informed written consent and follow the study procedures

Exclusion Criteria:

* Concurrent participation in any clinical trial or study
* With renal, liver or thyroid dysfunction, cognitive impairment, or any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study
* Multiple pregnancies
* Pre-existing DM
* With physical restriction that prevents from exercising
* Substance abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-06-28 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects developed GDM | 24-28 weeks gestation

SECONDARY OUTCOMES:
Proportion of neonates born with large for gestational age (LGA) | within 48 hours after delivery
Proportion of neonates born with macrosomia | within 48 hours after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Chan RS, Tam WH, Ho IC, Kwan MW, Li LS, Sea MM, Woo J. Randomized trial examining effectiveness of lifestyle intervention in reducing gestational diabetes in high risk Chinese pregnant women in Hong Kong. Sci Rep. 2018 Sep 14;8(1):13849. doi: 10.1038/s41598-018-32285-6. PMID 30218012